CLINICAL TRIAL: NCT06962631
Title: V-IMMUNE® for Immune Thrombocytopenia: A Prospective Multicenter Study to Evaluate the Efficacy and Safety of Human Immunoglobulin in Adult and Pediatric Participants With Immune Thrombocytopenia. TIP Study
Brief Title: V-IMMUNE® for Immune Thrombocytopenia
Acronym: TIP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: On Pharma Importadora, Exportadora e Distribuidora de Medicamentos LTDA. (Other)
Collaborators: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TIP study
Record Dates: First submitted 2025-04-15; First posted 2025-05-08 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-07

CONDITIONS: Immune Thrombocytopenia (ITP)
Keywords: phase III; clinical trial; immune thrombocytopenia; human immunoglobulin; platelets
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — V-Set Domain-Containing T-Cell Activation Inhibitor 1

STUDY DESIGN:
Intervention Model Description: All participants will get the same intervention: IV immunoglobulin for 2 consecutive days. Participants meeting the inclusion criteria will receive V-IMMUNE® at a dose of 1 g/kg once daily for two consecutive days, with infusion rates progressively increased to a maximum of 0.06 mL/kg/min, provided no adverse events occur. Pre-medication with intravenous normal saline and diphenhydramine is administered to mitigate infusion-related risks.
Masking Description: No mask is possible with this intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention arm (Experimental): Intervention arm will receive a human normal immunoglobulin to be administered intravenously, once daily for 2 consecutive days (Day 1 and Day 2).
  If the platelet count is not maintained for the desired duration after the first immunoglobin infusion, and at the discretion of the investigator and the patient/legal representative, participants may receive up to one additional cycle between Day 15 and Day 30 Pre-Medication Rapid IV infusion of 500 mL of 0.9% saline, 50 mg of diphenhydramine IV followed by saline 0.9% slow infusion Pediatrics, before the infusion of PSI, an IV infusion of 0.9% sodium chloride (normal saline) at 10 mL/kg over 1 hour, up to a maximum volume of 500 mL, will be administered, along with diphenhydramine 1.25 mg/kg IV, up to a maximum dose of 50 mg.
  At the end of the V IMMUNE® infusion, administer 0.9% sodium chloride IV at 10 mL/kg, up to a maximum of 500 mL, at an infusion rate of 10 mL/kg, to maintain a patent venous access for at least 30 to 40 minutes.
  Interventions: Biological: 5% (5g/100 ml) intravenous immunoglobin

INTERVENTIONS:
Biological: 5% (5g/100 ml) intravenous immunoglobin — A 5% human normal immunoglobulin I.P. (5 g/100 mL) V-IMMUNE® will be administered at a dose of 1 g/kg, intravenously, once daily for 2 consecutive days (Day 1 and Day 2). The infusion rate starts at 0.01 mL/kg/min during the first 30 minutes and is gradually increased up to 0.06 mL/kg/min if no adverse events occur. This will constitute the first cycle of V-IMMUNE® treatment. The dose of 1 g/kg/day on 2 consecutive days is consistent with recommendations for the use of other IVIG products in Immune Thrombocytopenia.
  If the platelet count is not maintained for the desired duration after the first V-IMMUNE® cycle, and at the discretion of the investigator and the patient/legal representative, participants may receive up to one additional cycle of V-IMMUNE®-at the same dosing regimen used in Cycle 1-between Day 15 and Day 30
  Pre-medication before infusion :
  IV rapidly infusion of 0.9% normal saline 500 mL, or 10 ml/kg pediatrics and diphenhydramine 50 mg IV or 1.25 mg/kg IV (pediatrics)
  Other Names: V-IMMUNE

SUMMARY:
This is a multicenter, prospective clinical trial evaluating the efficacy and safety of V-IMMUNE®, a 5% human normal immunoglobulin formulation administered intravenously, for the treatment of immune thrombocytopenia (ITP) in patients aged ≥1 year. The primary objective is to assess the proportion of patients achieving a platelet count ≥50,000/mm³ on or before Day 9 following the first infusion. The trial employs a single-group design, comparing outcomes to historical controls derived from the literature. Eligible patients must have a confirmed diagnosis of ITP with a platelet count ≤20,000/mm³ and no concurrent conditions likely to cause thrombocytopenia. Key exclusions include non-immune thrombocytopenia, active sepsis, pregnancy or lactation, hypersensitivity to blood products or IgG preparations, and various significant comorbidities (e.g., uncontrolled hypertension, severe hepatic or renal impairment, recent rituximab use). The intervention consists of V-IMMUNE® at a dose of 1 g/kg, administered once daily for two consecutive days, with infusion rates titrated from 0.01 mL/kg/min to 0.06 mL/kg/min. Standard pre-medication protocols (IV normal saline and diphenhydramine) are administered to mitigate infusion-related reactions and reduce the risk of thromboembolic events. Patients will be monitored at multiple time points from baseline through Day 90, with primary efficacy evaluation at Day 9. Secondary endpoints include duration of platelet response, overall treatment response rate, bleeding events, and incidence of infusion-related adverse events.

DETAILED DESCRIPTION:
TIP Study V-IMMUNE® for Immune Thrombocytopenia: A prospective multicenter study to evaluate the efficacy and safety of Human Immunoglobulin in adult and pediatric participants with immune thrombocytopenia.

Introduction Immune thrombocytopenia is an autoimmune disease characterized by thrombocytopenia (<100,000/mm³) and an increased risk of bleeding.

Antibody- and/or T-cell-mediated platelet destruction plays a key role in the pathophysiology of immune thrombocytopenia. Newly diagnosed immune thrombocytopenia is characterized by a platelet count <100,000/mm³ within three months of diagnosis. When remission is not achieved or the treatment response is not sustained within three to twelve months, it is considered persistent immune thrombocytopenia. When thrombocytopenia lasts for more than 12 months, it is considered chronic immune thrombocytopenia.

Bleeding in adults with immune thrombocytopenia can range from mild events, such as cutaneous petechiae, to potentially life-threatening events, such as organ bleeding and intracranial hemorrhage. The goal of treatment is to raise the platelet count to levels that can maintain hemostasis, preventing bleeding events or controlling any active bleeding. Hemorrhagic events are associated with worse outcomes and increased mortality in patients with chronic immune thrombocytopenia. Patients who required hospitalization due to bleeding had a 4.9-fold higher risk of mortality at 1 year and a 3.4-fold higher risk at 5 years compared to those who did not experience bleeding. Although most patients with immune thrombocytopenia present only with mild bleeding, the fear of more severe bleeding can negatively impact patients' quality of life. Therefore, experiencing a severe bleeding event is associated with a poor prognosis, increased risk of mortality, and may have substantial negative impacts on a patient's quality of life.

Treatment guidelines for immune thrombocytopenia in adults suggest maintaining platelet counts >20,000-30,000/mm³ in symptomatic patients, as the risk of severe bleeding increases below this threshold. In Brazil, the treatment guideline for immune thrombocytopenia in adults from the Brazilian Association of Hematology, Hemotherapy and Cellular Therapy (ABHH)/Guideline Project of the Brazilian Medical Association (AMB) recommends corticosteroids and intravenous immunoglobulin (IVIG) as first-line therapy for patients with platelet counts <30,000/mm³ and active bleeding. The combination of these therapies may be indicated in emergency situations.

The International Consensus for the treatment of immune thrombocytopenia in pediatrics also recommends observation in newly diagnosed patients without bleeding. Any severe bleeding (grade 4) requires immediate hospitalization for treatment to raise platelet levels until the bleeding subsides. Any moderate bleeding (grade 3) requires consideration for hospitalization and therapy. In cases of moderate or severe bleeding, IVIG and anti-D immunoglobulin (not approved in Brazil for immune thrombocytopenia) may be indicated.

The pediatric immune thrombocytopenia treatment guideline from the Brazilian Association of Hematology, Hemotherapy and Cellular Therapy (ABHH)/Guideline Project of the Brazilian Medical Association (AMB) recommends IVIG or corticosteroids as first-line therapy for newly diagnosed patients with platelet counts <20,000/mm³ and active bleeding.

In emergency situations, regardless of the phase of the child's immune thrombocytopenia, combined therapy with platelet transfusions, intravenous corticosteroids, and IVIG is indicated. Splenectomy may be considered when there is no response to corticosteroids or IVIG and the patient continues to have significant central nervous system bleeding. Thrombopoietin receptor agonists may also be considered.

IVIG acts in immune thrombocytopenia by blocking the mechanism of peripheral platelet destruction, which involves opsonization mediated by Fc fragments of antibody-coated platelets. The effect of IVIG is rapid, increasing the platelet count within 24 hours of administration. Platelet levels typically continue to rise over the next 24 to 48 hours. The original dose was 0.4 g/kg/day for up to 5 days; however, similar results are achieved with a dose of 1 g/kg/day given in 1 or 2 doses. In elderly patients or those with compromised cardiac or renal function, the lower dose may help prevent acute volume overload.

The availability of new products that demonstrate efficacy and safety for the treatment of immune thrombocytopenia is necessary. Therefore, it becomes essential to conduct this study to appropriately request registration from ANVISA (Brazilian Drug Agency) for the polyvalent human immunoglobulin for intravenous use (V-IMMUNE® ) produced by the Virchow laboratory in India, for potential use in Brazil

OBJECTIVES Primary Objective To evaluate the efficacy of the human normal immunoglobulin preparation V-IMMUNE® in improving platelet counts in patients with immune thrombocytopenia by or before Day 9 after the first infusion.

Secondary Objectives

* To determine the safety and tolerability of V-IMMUNE® at the dose used in this study;
* To determine the proportion of individuals with immune thrombocytopenia who achieve a complete or partial therapeutic response by or before Day 9 after the first dose of V-IMMUNE®;
* To determine whether V-IMMUNE® maintains platelet counts ≥ 50,000/mm³ in individuals with immune thrombocytopenia for a period similar to that of a historical control after the first treatment cycle;
* To compare the occurrence of bleeding in individuals with immune thrombocytopenia after the use of V-IMMUNE® with the results of historical controls.

METHODS Design A prospective, Phase III, open-label, non-randomized, multicenter, single-group study with a historical control, for intravenous administration of V-IMMUNE®.

Recruitment Plan Each participating center must identify and consecutively enroll potentially eligible patients. In case of doubt regarding the eligibility criteria, the center must immediately contact the sponsor's representative before enrolling the patient in the study.

Recruitment will occur through approximately 8 to 15 nationally recognized hematology centers specialized in the treatment of immune thrombocytopenia with intravenous immunoglobulin infusion.

Screening During the screening of potential participants, a standardized form will be used to confirm eligibility criteria. The investigator responsible for presenting the study must explain the protocol in detail to the patient and/or legal guardian/representative who, upon agreeing to participate and signing the Informed Consent Form (ICF), will be registered in the data collection system. Every screened participant who does not meet the inclusion criteria (screening failure) must be recorded along with the reason for non-inclusion.

Approach Patients who meet the inclusion criteria will be approached at the participating centers for enrollment in the TIP study. Once the Informed Consent Form (ICF) is signed, the participant will begin receiving V-Immune® On-Pharma according to the protocol.

Randomization Method and Maintenance of Allocation Concealment As this is a single-group study, there will be no randomization. Blinding As this is a single-group study in which eligible patients have a clinical/therapeutic indication for the use of immunoglobulin, blinding is not necessary.

Experimental Intervention The Investigational Product (IP) is V-IMMUNE®, normal human immunoglobulin I.P. 5% (5g/100 mL), manufactured from qualified human plasma for intravenous use. Each vial contains Human Immunoglobulin 50 g/L, Maltose 100 g/L, and Water for Injection. The 5% Human Immunoglobulin solution for intravenous administration I.P. is a sterile, pyrogen-free preparation of normal human immunoglobulin in a single-dose form for intravenous infusion. Each 10 mL, 50 mL, and 100 mL contains 0.5 g, 2.5 g, and 5 g of normal human immunoglobulin, respectively, and is prepared from qualified human plasma using membrane filtration, combined chromatographic steps, and viral inactivation procedures. The IgA content does not exceed 2 mg/mL. The IgG subclass distribution is similar to that found in normal human serum.

The manufacturing process uses plasma collected from donors who are screened based on medical history, in accordance with regulatory authority guidelines. The blood is tested for mandatory infectious diseases. Only plasma that tests negative for HBsAg, HCV, and HIV antibodies is used in the process.

Storage and Use Conditions of the IMP V-IMMUNE® immunoglobulin must be stored in a secure, access-restricted area, preferably in a refrigerator, protected from light, and maintained at a temperature of 2°C to 8°C. V-IMMUNE® immunoglobulin must not be frozen.

Administration Before use, all vials must be visually inspected for discoloration, particles, or fibers; if the contents of a vial are cloudy or contain particulate matter, it must not be used. V-IMMUNE® must not be shaken, frozen, or used if the solution has been frozen. The IMP should be at room temperature when infused.

Normal human immunoglobulin I.P 5% (5g/100 ml) V-IMMUNE® will be administered at a dose of 1 g/kg, intravenously, once daily for two consecutive days (Day 1 and Day 2). The infusion rate should start at 0.01 ml/kg/min for the first 30 minutes, increasing gradually to 0.06 ml/kg/min if no adverse events occur. This will constitute the first treatment cycle with V-IMMUNE®. The 1 g/kg/day dose for two consecutive days is consistent with recommendations for other IVIG products used in Immune Thrombocytopenia.

If the platelet count is not maintained for the desired duration after the first cycle of V-IMMUNE®, and at the discretion of the investigator and the participant/legal guardian, participants may receive one additional cycle of V-IMMUNE®, using the same dosing schedule as Cycle 1, between Day 15 and Day 30.

All infusions will be administered by trained personnel under the direct supervision of the principal investigator or a designated delegate.

V-IMMUNE® will be administered intravenously (via peripheral or central vein) through a dedicated infusion line. Mixing or administering any other product (including saline) with V-IMMUNE® is strictly prohibited.

If an adverse event (AE) occurs, the infusion should be interrupted for 20 to 30 minutes. The patient should be hydrated and given antihistamines, analgesics, and antiemetics. Once symptoms improve, the infusion may be resumed at a reduced rate, starting again at the initial infusion speed. Intolerance at any infusion rate must be recorded as an adverse event (AE) at that specific rate. If a participant experiences the same AE at the same rate twice and both events are recorded, further increases in infusion rate should not exceed the last tolerated speed. The patient will be observed for 60 minutes after the infusion ends for clinical evaluation and monitoring for potential adverse events.

In cases of clinically significant hypotension and/or anaphylactic reactions, in addition to stopping the infusion and administering appropriate supportive care as deemed necessary by the investigator (which may include epinephrine, antihistamines, corticosteroids, supplemental oxygen, volume expansion, etc.), these events must be documented in the source file and Case Report Form (CRF) as AEs. The participant may, at the investigator's discretion, be withdrawn from the study. In such cases, the participant may still choose to complete the follow-up visits.

For individuals at increased risk of thromboembolism (e.g., advanced age, obesity, hypertension, diabetes mellitus, history of thromboembolic events, known acquired or congenital thrombophilic disorders, prolonged immobilization, severe hypovolemia, hyperviscosity), the infusion rate should be kept as low as possible.

Pre-medication Prior to IMP Infusion In adult individuals, prior to IMP infusion, a rapid infusion of 500 ml of 0.9% sodium chloride (NaCl), IV, will be administered along with diphenhydramine 50 mg, IV. At the end of the V-IMMUNE® infusion, continue 0.9% NaCl, IV, at an infusion rate of 1 ml/kg/hour for at least 30 to 40 minutes.

In pediatric individuals, prior to IMP infusion, 0.9% NaCl IV will be administered at 10 ml/kg along with a maximum of 500 mL with diphenhydramine at 1.25 mg/kg over 1 hour with a maximum dose of 50 mg. At the end of the V-IMMUNE® infusion, continue 0.9% NaCl, IV, at an infusion rate of 10 ml/kg for at least 30 to 40 minutes with the maximum amount administered of 500 mL.

Pre-medication is necessary and is part of the routine protocol for infusion of these blood products. The rapid crystalloid infusion prior to administration reduces the risk of headache and aseptic meningitis following the infusion, as well as the risk of thromboembolic events. The crystalloid administration after the investigational product infusion is essential to reduce the risk of a severe and potentially fatal adverse event due to an anaphylactic episode, allowing for rapid intravenous medication management in a potentially shocked patient and avoiding the need for emergency central venous access.

Control Historical controls (literature data). No co-interventions are allowed.

Contraindications and Precautions Related to the IP Normal Human Immunoglobulin for Intravenous Administration I.P. 5% is contraindicated in patients with selective IgA deficiency.

Patients may experience severe hypersensitivity reactions or anaphylaxis in the presence of detectable IgA levels after infusion of Normal Human Immunoglobulin I.P. 5%. The occurrence of severe hypersensitivity reactions or anaphylaxis under such conditions should prompt consideration of alternative therapy.

The intravenous solution of Normal Human Immunoglobulin should only be administered intravenously.

Additional listed precautions regarding the use of Normal Human Immunoglobulin I.P. 5% include:

Hypersensitivity: Immediate hypersensitivity and anaphylactic reactions are rare but possible. If hypersensitivity occurs, immediately stop the infusion and initiate appropriate treatment. Medications such as epinephrine and antihistamines should be readily available for the immediate treatment of acute hypersensitivity reactions, including anaphylaxis.

Renal dysfunction: Acute renal failure, osmotic nephropathy, and death may occur with IVIG use. Ensure that the patient is not hypovolemic prior to administration. In patients at risk of renal dysfunction due to pre-existing renal insufficiency or predisposition to acute renal failure (e.g., diabetes mellitus, hypovolemia, obesity, use of nephrotoxic medications, or age >65), IVIG should be administered at the minimum infusion rate.

Aseptic Meningitis Syndrome (AMS): Rarely occurs with IVIG treatment. May begin within hours to 2 days after treatment. Discontinuation of IVIG usually leads to full recovery without sequelae. More common with high doses (2 g/kg) and/or rapid infusion.

Hemolysis: IVIG products may contain blood group antibodies that act as hemolysins, coating red blood cells and causing a positive direct antiglobulin test and, rarely, hemolysis. Delayed hemolytic anemia may occur due to red cell sequestration and acute hemolysis, consistent with intravascular hemolysis.

Transfusion-Related Acute Lung Injury (TRALI): Non-cardiogenic pulmonary edema may occur after IVIG administration. TRALI is characterized by severe respiratory distress, pulmonary edema, hypoxemia, normal left ventricular function, and fever, typically occurring 1 to 6 hours post-treatment. Patients should be monitored for pulmonary adverse events. If TRALI is suspected, appropriate tests should be conducted for anti-neutrophil antibodies in both the product and patient serum. Treatment includes oxygen therapy and ventilatory support.

Transmissible Agents: Normal Human Immunoglobulin I.P. 5% is derived from human plasma. Due to effective donor screening and manufacturing processes, the risk of viral disease transmission is extremely low. The theoretical risk of Creutzfeldt-Jakob disease (CJD) transmission is also considered extremely remote.

Monitoring - Laboratory Tests: Periodic monitoring of renal function and urine output is crucial in patients at increased risk of acute renal failure. Renal function (including serum urea and creatinine levels) should be assessed before the initial infusion and periodically as per the visit schedule. Due to a potentially increased risk of thrombosis, baseline blood viscosity assessment should be considered in patients at risk of hyperviscosity, including those with cryoglobulinemia, fasting chylomicronemia/markedly elevated triglycerides, or monoclonal gammopathies. If signs/symptoms of hemolysis are observed post-infusion, appropriate lab tests should be conducted. In cases of suspected TRALI, tests for anti-neutrophil antibodies should be performed on the product and patient serum.

Patient Information: Patients should be instructed to immediately report symptoms such as decreased urine output, sudden weight gain, fluid retention, edema, and/or shortness of breath-which may indicate kidney injury.

Pregnancy - Category C: Reproduction studies in animals have not been conducted with Normal Human Immunoglobulin for IV use. It is also unknown whether it can cause fetal harm when administered to a pregnant woman or affect reproductive capacity. It should be used during pregnancy only if absolutely necessary. Pregnant women are part of this study's exclusion criteria.

Presentation of the Investigational Product (IP) Normal human immunoglobulin for intravenous administration I.P. 5%, V-IMMUNE®, is available in vials of 0.5g/10 mL, 2.5g/50 mL, and 5g/100 mL (5% concentration), in single-dose format for intravenous administration.

IP Manufacturing and Labeling V-IMMUNE® immunoglobulin is manufactured, packaged, and labeled by Virchow Biotech Private Limited, and imported by OnPharma Importadora Exportadora e Distribuidora de Medicamentos LTDA, in accordance with current regulations. The preparation and labeling of the IP follow Good Manufacturing Practice (GMP) guidelines, and its distribution adheres to Good Distribution Practice (GDP) guidelines. IP labels will be in Portuguese and meet Brazilian legal requirements.

Follow-Up

Visits:

Day 1 and Day 2: IVIG infusion. Patients are assessed Before infusion; During infusion and up to 30 minutes after; At 1 hour, 24 hours, and 72 hours after the start of the investigational product infusion.8 Days 3, 5, 9, 15, 30, 90: Clinical and laboratory evaluations. Monitoring Real-time patient symptom diary as source documentation for AE collection. Laboratory

Day 1 (baseline data):

Complete blood count with platelet count (confirmed by peripheral blood smear), reticulocyte count, electrolytes, serum glucose, urea, creatinine, AST, ALT, LDH, total bilirubin, and urinalysis (type 1). Tests used to define inclusion and exclusion criteria must be collected at the participating center's certified laboratory after signing the informed consent/assent form, unless the patient already has results from the past 48 hours or from the same certified laboratory of the participating center.

Day 2 (±1 day):

platelet count (peripheral smear confirmation)

Day 3 (+ 1 day) and 5 (±1 day):

CBC with platelet count (peripheral smear confirmation), reticulocyte count, electrolytes, serum glucose, BUN, creatinine, AST, ALT, LDH, total bilirubin, urinalysis; Haptoglobin, direct Coombs test.

Days 9 (±1 day), 15 (±1 day), 30 (±2 days) e 90 (±5 days):

Platelet count (confirmed on a peripheral smear). Sample Size Calculation and Statistical Analysis Plan It is expected that 83% of patients will achieve a platelet count ≥50,000/mm³ on or before Day 9.12 For 80% power and a lower boundary of a one-sided 95% confidence interval (CI) ensuring at least a 60% response rate, using the normal approximation to the binomial distribution, a minimum of 31 patients must be studied, without allowing for losses to follow-up.

The study visits are identified as follows:

* Visit 1: screening, eligibility assessment, and first PSI infusion.
* Visit 2: second PSI infusion (24 hours after the start of the first V-IMMUNE® infusion, on consecutive days).
* Follow-up: 6 follow-up visits on Days 3, 5, 9, 15, 30, and 90.
* Study completion visit - Day 90: for all individuals, this visit will occur approximately 3 months after the first infusion of the last V-IMMUNE® cycle and will serve as the study completion visit for all participants.

A complete medical history will be obtained from each participant at the first visit. The history will include, specifically, documentation of the diagnosis of immune thrombocytopenia, the rationale for excluding other causes of non-immune thrombocytopenia, general medical history, prior use and/or reactions to any IVIG or other blood products, history and treatment of immune thrombocytopenia, and history of bleeding/hemorrhage.

The medical history should include, when relevant, the use of previous IVIG treatments; the product name, unit dose, and how well it was tolerated by the participant. Prior use of IVIG must be documented in the source documents and in the participant's CRF. Additionally, the treatment regimen and dose of corticosteroids, dapsone, azathioprine, cyclosporine A, danazol, vincristine sulfate, or mycophenolate mofetil, thrombopoietin receptor agonists, cyclophosphamide, and attenuated androgens must be documented in the source documents and in the participant's CRF, as well as any other chronic medications used within the previous 6 months.

All female individuals of childbearing potential will undergo a pregnancy test (human chorionic gonadotropin - hCG measurement) in blood, except in cases of documented impossibility of pregnancy (for example: hysterectomy, bilateral oophorectomy, or female children who have not yet reached menarche).

An interim analysis is planned after 6 months of study or once 50% of the sample size has been reached, whichever comes first

Special situations in case of participant's withdrawal:

1. Study participant becomes pregnant during participation in the study:

   Discontinue any further administration of PSI;
   * Participant's Clinical follow-up through routine care;
   * Participant will continue to be followed by the study;
   * Obtain informed consent from the pregnant participant to request authorization to monitor her pregnancy;
   * If authorized through a specific informed consent form, even after completing participation in the study, the investigator must contact the pregnant participant every three months to monitor the pregnancy.
   * The results of this follow-up must be entered into the CRF.
2. Female partner of a male study participant becomes pregnant during the study - No action is required regarding the study participation of the male participant; Obtain informed consent from the male participant's partner to request authorization to monitor her pregnancy; if authorized the investigator must contact the pregnant particpant

Strategies to Reduce Loss to Follow-Up and Manage Participation MISSED APPOINTMENTS AND/OR SCHEDULED COLLECTIONS

1. Reschedule the visit within the time frames described above. If the participant wishes to continue in the study but cannot attend on the proposed date, indicate in the CRF system that the participant "forgot/could not attend" and reschedule the next visit according to the timeline.
2. If the participant reports being unable to travel to the center: assess the possibility of a home visit/sample collection.

Loss to follow-up will only be considered if, at the end of the study, all attempts to contact the participant have failed and no data collection is possible.

REFUSAL TO PARTICIPATE IN SPECIFIC STUDY STAGES

1. Explain the importance of the study and the value of full participation;
2. If the participant no longer wishes to continue treatment, encourage them to at least attend the final laboratory collection and final consultation, and to accept phone contact for information on vital status, bleeding, and adverse events;
3. If the participant does not want to undergo all data collections, encourage them to at least attend the final consultation and accept phone contact for information on vital status, bleeding, and adverse events;
4. If the participant states they no longer wish to receive phone calls, online forms, emails, or attend the final visit, indicate "loss to follow-up" in the CRF system.

WITHDRAWAL OF CONSENT "Withdrawal of Consent" will be considered when the participant no longer wishes to undergo any study procedures. This right will be acknowledged to the participant through the Informed Consent Form (ICF). From the moment consent is withdrawn, no further study procedures will be conducted, and no new data will be collected. Data collected up to that point will remain in the study database; however, if the participant requests that they be removed, those data will no longer be used.

DATA QUALITY CONTROL Electronic System and Data Collection The data collection system for the TIP study is Clinical One - Oracle, a web-based platform available 24/7, with functionalities including patient registration, follow-up data entry, data cleaning, and export for statistical analysis.

Once qualified to participate in the TIP study, all centers will receive training on how to use the software, along with an operations manual.

Electronic case report forms must be accessed online via the study system. Data are entered by the site team, and all forms must be electronically signed by the site's principal investigator or designated personnel. Usage instructions will be made available to investigators.

Data Quality Assurance

Several procedures will ensure data quality, including:

All researchers will attend training sessions before study initiation to ensure procedural consistency, including data collection; Investigators will receive a detailed operations manual describing each protocol step; Investigators may contact the sponsor's representative to resolve any issues that may arise; Data entered into the study system undergo multiple validations, such as checks for blank fields, plausible and allowed value ranges, and logical checks. The system alerts the investigator of any issues at the time of entry; The sponsor's representative will periodically review data extracted from the system to assess completeness and identify inconsistencies. These findings will be shared with site teams for resolution via regular "queries"; Statistical techniques will be used periodically to detect possible fraud; 100% monitoring of data will be conducted at the sites during the study; The sponsor's representative will review monthly detailed reports on screening, enrollment, follow-up, data consistency, and completeness, and will act immediately on any problems.

Site Monitoring Monitors will visit all participating centers to ensure protocol adherence and compliance with good clinical practice. Visits will follow a monitoring plan to ensure participant safety and proper data collection. Frequency will depend on recruitment rates, with more frequent visits to high-enrolling centers or those with outstanding issues. Training sessions will be organized at study start and as needed thereafter.

All information during monitoring visits will be treated with strict confidentiality. Upon sponsor request, investigators must grant direct access to all trial-related records.

Source Data and Records Source data are defined as all information related to clinical findings, observations, or other study activities recorded in original documents or certified copies. The investigator will permit study-related monitoring, audits, ethics committee reviews, and regulatory inspections with direct access to source data/records.

Protocol Adherence This protocol outlines study objectives, required procedures, and data to be collected. Under no circumstance is a researcher authorized to collect additional data or perform extra procedures related to the investigational product beyond the study's intent. If incidental data are collected, the investigator must report them to the sponsor and refrain from using them for any purpose outside the study, except for appropriate participant monitoring.

Significant deviations from protocol procedures or criteria are considered violations, potentially compromising data integrity, result validity, or participant safety. Protocol violations require formal reporting and corrective actions.

Study Approval The study will be submitted to a Research Ethics Committee (REC) as per regulations and will only begin after protocol approval. It has also been submitted for review and oversight by the Brazilian Health Regulatory Agency (Anvisa), according to Law No. 14.874/2024 and Anvisa RDC No. 204/2017.

International Guidelines The study will follow the Good Clinical Practice (GCP) guidelines of the International Council for Harmonisation (ICH E6/R3).

Brazilian Regulations

This protocol was developed and will be conducted in compliance with the following:

1. Law No. 14.874/2024;
2. CNS Resolution No. 466/12;
3. Anvisa RDC No. 945/2024;
4. Operational Standard No. 001/13;
5. Other relevant regulations. Informed Consent or Assent The Informed Consent Form (ICF) was written using lay, understandable language, without technical terms or foreign expressions. Consent will be obtained in a private, quiet environment by the investigator or a formally delegated team member. They will explain the study details, procedures, risks, and potential benefits. Once it's confirmed that the participant/legal guardian has no further questions, they will be given time to read and discuss the ICF before deciding. It must be emphasized that participation is entirely voluntary, and refusal will not affect care.

If consent is granted, the ICF will be signed and dated by the participant or legal representative and by the investigator/delegate, in two copies-one for the center's files and one for the participant. The center's copy will be securely stored with restricted access. ICFs will be retained for 5 years after study completion.

Maintenance and Archiving of Data and Documents The principal investigator must maintain a study archive with all documents (source documents) on-site for 5 years. If the investigator leaves the institution, documentation must be transferred to their successor, and the sponsor must be notified of this change. The principal investigator is also responsible for periodically updating the Delegation of Duties Log for the research team.

Data Confidentiality The principal investigator must maintain all study documents on-site for 5 years. If they leave the institution, documents must be handed over to their replacement. The sponsor must be informed of researcher departures and new appointments. The principal investigator must also regularly update the Delegation of Duties Log.

Risks and Benefits Risks to participants involve both the intervention and data collection. Adverse events (AEs) related to the intervention are listed in Section 3.7.1.2. Risks will be minimized by following the manufacturer's guidelines, clinical evaluation, and routine premedication. Participants will be advised to contact the study team if AEs occur.

Blood sampling may cause local pain, bruising, or phlebitis. These will be minimized by using trained healthcare professionals.

There is a risk of confidentiality breaches in data collection. To minimize this, all records will be confidential and accessed only by study personnel. Participant identities will be replaced with a study ID number.

As for benefits, participants are expected to experience increased platelet levels, reducing the risk of clinically significant bleeding. The study may also benefit others with immune thrombocytopenia by providing a potential new therapeutic option.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥1 year;
* Confirmed diagnosis of immune thrombocytopenia ( newly diagnosed, persistent or chronic);
* Platelet count ≤20,000/mm³ at the time of enrollment;
* No other conditions that, in the investigator's opinion, could cause thrombocytopenia;
* Agreement to use effective contraceptive practices/methods throughout the entire study participation by female patients of childbearing potential and able to become pregnant, unless there is a documented medical contraindication.

Exclusion Criteria:

* Non-immune thrombocytopenia
* Active sepsis
* Pregnancy (pregnant or breastfeeding)
* History of hypersensitivity reaction to blood or blood products, IVIG, or any other IgG preparation
* Intolerance to any component of V-IMMUNE®
* Previous diagnosis of IgA deficiency, history of reactions to products containing IgA, or history of anti-IgA antibodies
* Participation in any other study involving an investigational product
* Known HIV, HCV, or HBV infection
* AST (TGO) and/or ALT (TGP) >2.5× the upper limit of normal or 2.5 times baseline values
* Serum creatinine >2× the upper limit of normal or 2 times baseline values
* BUN >2.5× the upper limit of normal or 2.5 times baseline values
* History of NYHA class III or IV heart failure
* Uncontrolled hypertension with systolic BP >180 mmHg or diastolic BP >100 mmHg
* A history of hyperviscosity states, transient ischemic attack (TIA), stroke, other thromboembolic events, or acute coronary syndrome (ACS)
* Neoplasia under active treatment
* Child-Pugh class B or C liver failure
* Alcohol, opioid, or psychotropic substance abuse within the past 12 months
* Receipt of rituximab within 6 months prior to Day 1
* Acute or chronic conditions (e.g., but not limited to, renal disease or diseases predisposing to renal impairment, coronary artery disease, or protein-losing enteropathy) that, in the investigator's opinion, may interfere with the conduct of the study

An acquired health condition such as chronic lymphocytic leukemia, multiple myeloma, or chronic or recurrent neutropenia (absolute neutrophil count <1,000/mm³)

History of hemolytic anemia

Receipt of any IV immunoglobin preparation within 1 month prior to Day 1

Use of corticosteroids, cyclophosphamide, azathioprine, or attenuated androgens with a planned dose increase before Day 10 following IV immunoglobin infusion

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2026-08-27 (Estimated); Study Completion 2027-02-27 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving a platelet count ≥50,000/mm³ on or before Day 9 following the first infusion | 9 days
  Evaluate the efficacy of V-IMMUNE® in raising the platelet count of individuals with immune thrombocytopenia to a threshold of 50,000/mm³ or greater by or before Day 9 following the first dose. The proportion will be the ratio between the number of patients who achieved platelet count ≥ 50,000/mm3 / total of patients who received at least one dose of V-Immune® and had laboratory assessments performed at least once during the scheduled visits within 9 days.

SECONDARY OUTCOMES:
Therapeutic response defined as the increase in platelets count | 9 days
  Proportion of individuals with immune thrombocytopenia who achieve a complete or partial therapeutic response by or before Day 9 following the first dose of V-IMMUNE®. Response criteria can be:
  1. Complete response (remission): platelet count ≥100,000/mm³ with no clinically significant bleeding;
  2. Partial response (remission): platelet count between 30,000-100,000/mm³ or at least double the baseline count, with no clinically significant bleeding.
Bleeding occurrence classified according to CTCAE version 5.0 | 30 days
  Number of bleeding events (as classified by the Common Terminology Criteria for Adverse Events [CTCAE], version 5.0; up to Day 30 after the first infusion.
Number of days with platelets count ≥ 50,000/mm3 | 90 days
  Duration (in days) during which the platelet count remains ≥50,000/mm³ following the first treatment cycle with V-IMMUNE®.
Proportion of infusions during which one or more adverse events (AEs) occurred | 72 hours
  Proportion of infusions during which one or more adverse events (AEs) occurred within a predefined temporal window post-infusion
Total number of adverse events infusion related during the whole study | 30 days
  Cumulative number of adverse events (AEs) occurring intra-infusion or within 72 hours post-infusion
Mean number of temporally associated adverse events (AEs) per infusion | 30 days
  Mean number of temporally associated adverse events (AEs) per infusion, calculated as the ratio of i/ii:
  i. the total number of AEs occurring during or within 72 hours of an infusion; ii. the total number of infusions.
Proportion of patients who experienced one or more adverse events (AEs) | 90 days
  Proportion of patients who experienced one or more adverse events (AEs) at any time during the clinical study. (total number of patients with at least one AE/ total number of patients)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Regina Loggetto, PhD, Principal Investigator — HCor Research Institute; Israel Silva Maia, PhD, Study Director — HCor research institute
Locations (2):
- Brazil (2):
  - IMIP Instituto de Medicina Integral Professor Fernando Figueira, Recife, Pernambuco
  - Santa Casa de Misericórida de São Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No
Due to the regulatory nature of this clinical trial-specifically aimed at obtaining market authorization for V-IMMUNE® in Brazil for patients with immune thrombocytopenia-we will not be able to share individual participant data (IPD) outside of the study team. All participant information is considered proprietary and confidential as part of the registration dossier being submitted to the Brazilian health authority. The study protocol, data collection, and analyses must remain under restricted access to fulfill legal, regulatory, and institutional requirements, which include protecting patient privacy and maintaining data integrity for the product's approval process. Consequently, no external IPD sharing is planned at this time.

REFERENCES:
- [Background] Goudouris ES, Rego Silva AM, Ouricuri AL, Grumach AS, Condino-Neto A, Costa-Carvalho BT, Prando CC, Kokron CM, Vasconcelos DM, Tavares FS, Silva Segundo GR, Barreto IC, Dorna MB, Barros MA, Forte WCN. II Brazilian Consensus on the use of human immunoglobulin in patients with primary immunodeficiencies. Einstein (Sao Paulo). 2017;15(1):1-16. doi: 10.1590/S1679-45082017AE3844. PMID 28444082
- [Background] Perez EE, Orange JS, Bonilla F, Chinen J, Chinn IK, Dorsey M, El-Gamal Y, Harville TO, Hossny E, Mazer B, Nelson R, Secord E, Jordan SC, Stiehm ER, Vo AA, Ballow M. Update on the use of immunoglobulin in human disease: A review of evidence. J Allergy Clin Immunol. 2017 Mar;139(3S):S1-S46. doi: 10.1016/j.jaci.2016.09.023. Epub 2016 Dec 29. PMID 28041678
- [Background] Buckley RH, Schiff RI. The use of intravenous immune globulin in immunodeficiency diseases. N Engl J Med. 1991 Jul 11;325(2):110-7. doi: 10.1056/NEJM199107113250207. No abstract available. PMID 2052044
- See also: Sponsor´s website — https://onpharma.com.br/